CLINICAL TRIAL: NCT06888960
Title: An Exploratory Clinical Study on the Safety of CC312 in Treating Patients With Refractory Autoimmune Diseases
Brief Title: Safety Study of CC312 in Autoimmune Disease Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: CytoCares Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC312-I-001
Record Dates: First submitted 2025-01-20; First posted 2025-03-21 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Systemic Lupus Erythematosus (SLE); Idiopathic Inflammatory Myopathy (IIM); Systemic Sclerosis (SSc); Rheumatoid Arthritis (RA); Primary Immune Thrombocytopenia (ITP); Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Myositis; Scleroderma, Systemic; Arthritis, Rheumatoid; Purpura, Thrombocytopenic, Idiopathic; Anemia, Hemolytic, Autoimmune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CC312 (Experimental): The patient received CC312 via intravenous administration.
  Interventions: Biological: CC312

INTERVENTIONS:
Biological: CC312 — After a 28-day screening period, subjects who meet the inclusion and exclusion criteria will be enrolled for baseline assessments and biological sample collection prior to the guided administration period. The guided dose of CC312 will be administered via IV infusion on Day -3, followed by safety and tolerability assessments on the third day after the initial administration (i.e., Day -1). The therapeutic dose of CC312 will be administered via IV infusion on Day 1, with subsequent infusions scheduled on Day 4, Day 8, Day 11, Day 15, Day 18, Day 22, and Day 25. Comprehensive safety and tolerability assessments will be conducted at each of these time points.

SUMMARY:
This study is an open-label, multiple-dose escalation, Investigator-Initiated Trial (IIT) clinical trial designed to evaluate the safety and tolerability of CC312 in adult patients with relapsed and refractory autoimmune diseases. The trial also assesses pharmacokinetics (PK) and preliminary efficacy.

CC312 is a trispecific T cell engager (TriTE) that targets the B cell surface antigen CD19, the T cell antigen CD3, and the T cell co-stimulatory molecule CD28. Given its mechanism of action, which is similar to the "biopharmaceutical version" of CAR-T, there is a higher risk of cytokine release syndrome (CRS) at the onset of infusion administration. Therefore, a lower priming dose will be administered before the therapeutic dosing phase to mitigate this risk and ensure safety, followed by a therapeutic dose to achieve and maintain efficacy.

The study is divided into three dose groups, with 3-6 subjects enrolled in each group, resulting in a total of 9-18 subjects in the study. A "3+3" dose escalation design is employed to systematically evaluate the safety and determine the optimal dose of CC312.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who fully understand the objectives, nature, methods of the study, and possible adverse reactions, voluntarily participate as subjects, and sign the informed consent form (ICF).
* Age ≥18 years (inclusive, based on the time of signing ICF), male or female.
* For SLE:

  1. Subjects who are diagnosed with SLE according to the 2019 European League Against Rheumatism (EULAR)/1997 American College of Rheumatology (ACR) diagnostic classification criteria;
  2. SLEDAI-2000 score of ≥ 8 points and at least one BILAG grade A or two BILAG grade B under standard treatment conditions;
  3. Meet one of the following conditions: antinuclear antibody (ANA) determined to be positive during the screening period, or anti-dsDNA antibodies higher than normal levels at screening, or anti-Sm antibodies higher than normal levels at screening;
  4. Before the first dose of the investigational drug, subjects must have received at least one of the following standard treatments for 12 weeks, and the dose must have been stable for at least 30 days (dose reduction is allowed and dose increase is not allowed ). Standard treatment regimen refers to the stable use of any of the following (alone or in combination): a. Antimalarial (hydroxychloroquine) monotherapy; b. Antimalarials in combination with oral corticosteroids (OCS, e.g., prednisone or other hormones at equivalent doses) and/or immunosuppressants (including mycophenolate mofetil, cyclophosphamide, leflunomide, methotrexate, tacrolimus, ciclosporin, azathioprine, Tripterygium wilfordii); c. OCS and/or immunosuppressant combination therapy. If the subject is receiving OCS (e.g., prednisone or other hormones at equivalent doses), the following criteria must be met: at screening and during the screening period, the maximum dose of OCS is 30 mg/day of prednisone (or other hormones at equivalent doses); other drugs and traditional Chinese medicines that affect immunity may be continued at the discretion of the investigator.
* For IIM:

  1. According to the 2017 EULAR/ACR Classification Criteria, diagnosed as possible or definite IIM-possible IIM: with a score of 5.5 points without biopsy; definite IIM: with a score of 6.7 points with biopsy;
  2. Meeting one of the following criteria: During or before the screening period, confirmed to have at least one positive myositis-specific autoantibody (MSA), myositis-associated autoantibody (MAA), or ANA;
  3. Conventional treatment is ineffective or the disease relapses after remission. Conventional treatment is defined as: the use of glucocorticoids (prednisone >1 mg/kg/d or equivalent dose) and/or at least one immunomodulatory drug: such as antimalarial drugs, azathioprine, mycophenolate mofetil, cyclophosphamide, methotrexate, tacrolimus, ciclosporin, and/or biological drug products: such as rituximab and belimumab.
* For IIM:

  1. Subjects who are diagnosed with SSc according to the 2013 EULAR/ACR diagnostic classification criteria;
  2. Meets one of the following criteria: positive ANA confirmed during or before the screening period, or at least one positive SSc-related antibody profile (such as Scl70, Th/To, RP11/12, U3RNP autoantibodies);
  3. Conventional treatment is ineffective or the disease relapses after remission. Conventional treatment is defined as: using glucocorticoids (prednisone > 0.5 mg/kg/d or equivalent dose) and cyclophosphamide, and any of the following immunomodulatory drugs: such as antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, ciclosporin, and/or biological agents: such as rituximab and belimumab, with a cumulative treatment duration > 6 months.
* For RA:

  1. Diagnosed with RA according to the 2010 EULAR/ACR diagnostic classification criteria;
  2. Disease Activity Score DAS28-ESR >3.2 (i.e., moderate activity or higher) during the screening period;
  3. Failure after treatment with at least one conventional disease-modifying antirheumatic drug (DMARD) and/or at least one targeted synthetic DMARD (tsDMARD)/biologic DMARD (bDMARD) (defined as no remission after at least 3 months of treatment);
  4. At screening, if the subject is taking prednisone or an equivalent dose of a glucocorticoid, the dose must be ≤10 mg/day and stable for at least 4 weeks before the first dose;
  5. The subject must have discontinued traditional Chinese medicine for the treatment of RA for ≥4 weeks before the first dose;
  6. Other DMARDs, except for methotrexate (MTX) (subjects who have been on routine MTX treatment for 12 weeks before enrollment, with a stable MTX dose for 4 weeks before enrollment), must meet the washout period requirements: discontinuation of conventional synthetic DMARDs (csDMARDs) (including but not limited to sulfasalazine, leflunomide, penicillamine, azathioprine, ciclosporin A, cyclophosphamide, hydroxychloroquine, etc.) and herbal agents (including Tripterygium wilfordii, total glucosides of paeony, sinomenine, etc.) for 4 weeks before the first dose; discontinuation of intra-articular, intramuscular, or intravenous corticosteroids for 4 weeks before the first dose; discontinuation of anakinra and etanercept for 4 weeks before the first dose; discontinuation of adalimumab and infliximab for 8 weeks before the first dose; discontinuation of golimumab, certolizumab pegol, and tocilizumab for 10 weeks before the first dose; discontinuation of abatacept for 12 weeks before the first dose; in addition, stable doses of nonsteroidal anti-inflammatory drugs (NSAIDs) are permitted to be continued.
* For ITP:

  1. Diagnosed with ITP according to the diagnostic criteria of the Chinese Guideline on the Diagnosis and Management of Adult Primary Immune Thrombocytopenia (2020 Edition);
  2. Ineffective response or relapse after at least one prior treatment regimen (including but not limited to TPO mimetics/agonists, corticosteroids, immunoglobulins, azathioprine, cyclophosphamide, and/or rituximab);
  3. At least 2 platelet count measurements (with an interval of more than 24 hours) from the screening period to before the first dose, with an average platelet count <30×109/Land no single platelet count>35×109/L;
  4. If receiving standard background therapy for ITP, the dose and frequency of this therapy should be stable for at least 4 weeks (dose change ≤10%) before the first dose.
* For AIHA:

  1. Diagnosed with AIHA according to the diagnostic criteria of the Chinese Guideline on the Diagnosis and Management of Autoimmune Haemolytic Anaemia (2022 Edition);
  2. Poor response after at least first-line treatment (corticosteroids);
  3. Presence of anaemia-related symptoms during the screening period;
  4. The dose of supportive care must be stable for at least 4 weeks before the first dose.
* Laboratory test results:

Complete blood count:

1. SLE, SSc, and IIM: Absolute neutrophil count ≥1.0 x109/L, haemoglobin ≥60 g/L, platelets ≥50 x109/L;
2. RA: Neutrophil count ≥1.5 x109/L, haemoglobin ≥90 g/L, platelets ≥100 x109/L;
3. ITP: Absolute neutrophil count ≥1.0 x109/L, haemoglobin ≥70 g/L, platelets ≥10 x109/L;
4. AIHA: Absolute neutrophil count ≥1.0 x109/L, platelets ≥50 x109/L (≥10 x109/L for patients with Evans syndrome and transfusion is permitted).

Liver function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <3 times the upper limit of normal (ULN), and total serum bilirubin ≤1.5×ULN (≤3.0×ULN for Gilbert's syndrome) or if bilirubin abnormality is caused by the study disease, participation is allowed upon investigator's judgment.

Renal function: For RA, ITP, and AIHA: Serum creatinine ≤1.5 times ULN, or calculated creatinine clearance >50 mL/min (Cockcroft-Gault formula).

* Left ventricular ejection fraction (LVEF) ≥50%.
* Female subjects of childbearing potential must agree to use effective contraception from the screening period until 6 months after the last dose. Additionally, they must agree to refrain from collecting or donating eggs during this period; any male partners of reproductive potential must also agree to use effective contraceptive measures during this period.
* Male subjects with reproductive potential must agree to use effective contraception from the screening period to 6 months after the last dose, and have no plans for reproduction or sperm donation. During this period, their female partners of childbearing potential must also agree to use effective contraception.

Exclusion Criteria:

* Subjects who have severe lupus nephritis (defined as urinary protein >6 g/24 h or serum creatinine >2.5 mg/dL or 221 μmol/L), or required treatment of active nephritis with protocol-prohibited drugs, or required hemodialysis or received prednisone ≥100 mg/d or equivalent glucocorticoid therapy for ≥14 days within 8 weeks before screening.
* Subjects who have central nervous system diseases caused by SLE or not caused by SLE within 8 weeks before screening (including but not limited to epilepsy, psychosis, posterior reversible encephalopathy syndrome, cerebrovascular accident, encephalitis, central nervous system vasculitis, etc.).
* Other types of IIM: inclusion body myositis, diabetic amyotrophy, juvenile myositis; severe muscle injury or myositis causing permanent weakness or cardiac involvement due to non-IIM causes (e.g., stroke).
* Pulmonary arterial hypertension associated with SSc requiring treatment; or rapidly progressive SSc-related lower gastrointestinal tract (small and large intestine) involvement (requiring parenteral nutrition), active antral vascular ectasia; previous renal crisis caused by SSc.
* Significant organ transplantation (e.g., heart, lung, kidney, liver) or history of hematopoietic stem cell/bone marrow transplantation.
* Concomitant presence of two or more immune diseases requiring systemic treatment, if the investigator deems the subject unsuitable for enrollment.
* IgA deficiency (serum IgA level <10 mg/dL).
* Have participated in any other clinical trials (including cell or gene therapy) within 4 weeks before screening or within 5 half-lives of the investigational product (whichever is longer).
* Have received CAR-T therapy within 6 months before screening.
* Have received B-cell depleting drug rituximab or equivalent treatments (targeting CD19, CD20, BAFF, etc.) within 1 month before screening, unless it can be demonstrated that B cells have returned to pre-treatment levels or within the normal range.
* Have received anti-SLE treatments (e.g., Saphnelo) other than standard therapy within 3 months before screening or within 5 half-lives of the investigational product (whichever is longer).
* Have received a live/attenuated vaccine within 4 weeks before screening or plans to receive a live/attenuated vaccine during the study.
* Active infection.
* History of Grade 3-4 (CTCAE v5.0) allergic reaction to another monoclonal antibody treatment, or known allergy to any component or excipient of the CC312 drug product (including recombinant proteins, polysorbate 80, etc.); patients with a ≤Grade 3 allergy lasting <24h may participate in this study after discussion with the investigator.
* Acknowledgement of or evidence of illicit drug use, drug abuse, or alcoholism.
* Subjects who have received major surgery within 4 weeks before screening or minor surgery within 2 weeks; wounds must be completely healed (surgical procedures such as catheter placement are not exclusion criteria).
* History of any of the following cardiovascular diseases within 6 months before screening: NYHA Class III or IV heart failure, myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmia, any ventricular arrhythmia, or other clinically significant heart disease.
* Any other serious underlying diseases (e.g., active gastric ulcer, uncontrolled seizures, cerebrovascular events, gastrointestinal bleeding, severe signs and symptoms of coagulation dysfunction, heart diseases), mental illnesses, psychological, familial, or endemic diseases that, in the investigator's judgment, may interfere with the planned staging, treatment, and follow-up; affect subjects; compliance; or expose the subjects to a higher risk of complications.
* Evidence of concurrent malignant tumors within less than 5 years before screening, excluding adequately treated cervical carcinoma in situ, localized cutaneous squamous cell carcinoma, basal cell carcinoma, localized prostate cancer, ductal carcinoma in situ of the breast, or urothelial carcinoma of stage ≤T1. Subjects with prostate cancer undergoing active surveillance are eligible for this study.
* Pregnant or breastfeeding women.
* Subjects with positive results for viral serological tests during the screening period: positive for human immunodeficiency virus antibody (HIV-Ab), hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV-Ab), or Treponema pallidum antibody (TP-Ab).
* Subjects with active or latent tuberculosis (positive T-SPOT) identified during the screening period.
* History of splenectomy treatment within 6 months prior to screening.
* ITP subjects: 1) Secondary immune thrombocytopenia secondary to SLE, chronic lymphocytic leukemia (CLL), immunodeficiency common variable (CVID), or antiphospholipid syndrome (APS); 2) Drug-induced thrombocytopenia; 3) Any bleeding event requiring treatment within 4 weeks prior to screening; 4) Within 2 weeks prior to screening, the subject has continuously used drug therapy that affects platelet function (including but not limited to aspirin, aspirin-containing compounds, clopidogrel, salicylates, and/or NSAIDs) for >3 days; 5) History of any arterial or venous thrombosis (stroke, transient ischaemic attack, myocardial infarction, deep vein thrombosis, or pulmonary embolism), or clinical symptoms and medical history suggestive of thrombophilia; or any of the following: known arrhythmia that increases the risk of thrombotic events (e.g., atrial fibrillation), or corrected QT interval (QTc) >450 msec; or a history of other coagulation abnormalities.
* ITP and AIHA subjects: Abnormal prothrombin time (PT), international normalized ratio (INR), and activated partial thromboplastin time (aPTT) that are considered clinically significant by the investigator.
* Other subjects whom the investigator judges to be unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-11-08 (Estimated); Study Completion 2026-11-08 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | 2 years
  Hematological DLT is defined as a Grade 4 toxic reaction (excluding lymphopenia) that is not attributable to the underlying disease and persists for more than 29 days.
  Non-hematological DLT refers to any Grade ≥4 toxicities that may be associated with CC312 treatment, or Grade 3 toxicities that may be associated with CC312 treatment and persist for ≥7 days during the DLT observation period following CC312 infusion.
Adverse events (AE)/serious adverse events (SAE) | 2 years
  All adverse events will be evaluated and graded according to the severity criteria of CTCAE (Common Terminology Criteria for Adverse Events) version 5.0, with the exception of Cytokine Release Syndrome (CRS) and Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS), which will be assessed using the ASTCT (American Society for Transplantation and Cellular Therapy) standard.

SECONDARY OUTCOMES:
Maximum Serum Concentration (Cmax) of CC312 | 2 years
  Blood samples will be collected for serum concentration analysis at the following time points: within 1 hour before (0 hour) and 1 hour after the infusion of the initial dose; within 1 hour before (0 hour) and 1 hour after the infusion of the first and second doses in the first and third weeks of the therapeutic dose; within 1 hour before (0 hour) and 1 hour after the infusion of the first dose in the second and fourth weeks of the therapeutic dose; and at the time of early withdrawal/end of study (EOS).
Area Under the Concentration-time Curve (AUC) of CC312 | 2 years
  The area under the concentration-time curve (AUC) over the dosing interval of 72 hours was calculated using the linear trapezoidal rule.
Minimum Concentration (Cmin) of CC312 | 2 years
  The timing of blood sample collection is consistent with the sampling time for Cmax determination.
Counts of peripheral B cells | 2 years
  Blood samples will be collected for CD19+ and CD20+ B cell subsets analysis:
  For the priming dose: within 1 hour before (0 hour) and at 1 hour and 24 hours after infusion.
  For the therapeutic dose in the first week: within 1 hour before (0 hour) and at 1 hour and 24 hours after the first and second doses.
  At early withdrawal/End of Study (EOS).
Cytokine Indicators | 2 years
  Including but not limited to IL-2, IL-6, IL-10, IFN-γ, TNF-α, etc.
Anti-drug Antibodies | 2 years
  Collect blood samples at specific time points for the analysis of anti-drug antibody (ADA) levels and neutralizing antibody (NAb) levels.
Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2000) score | 2 years
  SLEDAI-2000 score is used to evaluate the clinical symptoms and disease activity of SLE. The score ranges from 0 to 15, with higher scores indicating more severe disease activity.
Total Improvement Score (TIS) | 2 years
  The Total Improvement Score (TIS) for idiopathic inflammatory myopathies (IIM) is a validated composite endpoint (typically ranging from 0 to 100) that quantifies the magnitude of overall clinical improvement, with higher scores denoting greater response and lower baseline scores often reflecting more severe disease activity.
ACR 20/50 score | 2 years
  ACR20/50 scores are standardized measures of treatment response in rheumatoid arthritis (RA) that directly correlate with reductions in disease activity. ACR20 represents the minimum clinically meaningful response in RA, while ACR50 indicates a robust response that is strongly associated with significant reduction in disease activity and improved long-term outcomes.
Overall Response Rate (ORR) for primary immune thrombocytopenia (ITP) | 2 years
  Overall Response Rate (ORR): proportion of ITP subjects whose efficacy is assessed as Complete Response (CR) or Response (R) at 4/8/12 weeks after the first infusion (treatment dose).
Overall Response Rate (ORR) for Autoimmune Haemolytic Anaemia (AIHA) | 2 years
  Overall Response Rate (ORR): proportion of subjects whose efficacy is assessed as CR or R at 4/8/12 weeks after the first infusion (treatment dose).
Peripheral blood mononuclear cell (PBMC) transcriptome analysis | 2 years
  Collect peripheral blood at baseline and specific post-treatment time points, isolate peripheral blood mononuclear cells (PBMCs), and decode the global gene expression profiles of immune cells.
Single-cell RNA sequencing (scRNA-seq) of peripheral blood mononuclear cells (PBMCs) | 2 years
  Peripheral blood is collected at baseline and specific post-treatment time points, followed by PBMC isolation and single-cell sequencing to resolve immune cell heterogeneity, uncover dynamic changes in cell states, and decipher cell-cell communication mechanisms.
Bone Marrow Lymphocyte Subtype Analysis | 2 years
  Collect bone marrow samples at baseline and specific post-treatment time points to analyze the proportion and counts of each immune cell subsets.
B-cell depletion analysis in lymph nodes | 2 years
  To evaluate the drug-induced deep depletion of B cells, lymph node samples are collected at baseline and specific post-dose time points to quantify the percentage and count of B cells within the tissue.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, China, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murimi-Worstell IB, Lin DH, Kan H, Tierce J, Wang X, Nab H, Desta B, Alexander GC, Hammond ER. Healthcare Utilization and Costs of Systemic Lupus Erythematosus by Disease Severity in the United States. J Rheumatol. 2021 Mar;48(3):385-393. doi: 10.3899/jrheum.191187. Epub 2020 Jul 1. PMID 32611669
- [Background] Fortuna G, Brennan MT. Systemic lupus erythematosus: epidemiology, pathophysiology, manifestations, and management. Dent Clin North Am. 2013 Oct;57(4):631-55. doi: 10.1016/j.cden.2013.06.003. PMID 24034070
- [Background] Cooper GS, Bynum ML, Somers EC. Recent insights in the epidemiology of autoimmune diseases: improved prevalence estimates and understanding of clustering of diseases. J Autoimmun. 2009 Nov-Dec;33(3-4):197-207. doi: 10.1016/j.jaut.2009.09.008. Epub 2009 Oct 9. PMID 19819109